CLINICAL TRIAL: NCT04191954
Title: Fasudil Eye Drop in Retinopathy Of Prematurity, Retinal Vascularization Induction and Disease Progression Inhibition, a Randomized Clinical Trial
Brief Title: Fasudil Eye Drop in Retinopathy Of Prematurity(ROP)
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zahra Rabbani Khah, Head of ophthalmic research center, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9800
Record Dates: First submitted 2019-11-29; First posted 2019-12-10 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-11

CONDITIONS: Retinopathy of Prematurity
MeSH Terms: conditions — Retinopathy of Prematurity

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fasudil eye drops (concentration 0.5 percent) (Active Comparator): twice daily
  Interventions: Drug: Fasudil eye drops (concentration 0.5 percent)
- receive artificial tears drop with the same frequency (Placebo Comparator)
  Interventions: Drug: receive artificial tears drop

INTERVENTIONS:
Drug: Fasudil eye drops (concentration 0.5 percent) — receive Fasudil eye drops (concentration 0.5 percent) twice daily
  Arms: Fasudil eye drops (concentration 0.5 percent)
Drug: receive artificial tears drop — receive artificial tears drop with the same frequency
  Arms: receive artificial tears drop with the same frequency

SUMMARY:
Eligible eyes are randomly assigned into two groups. Group A receive Fasudil eye drops (concentration 0.5 percent) twice daily. Group B, receive artificial tears drop with the same frequency. Retinal specialists who are expert in Retinopathy Of Prematurity field will perform fundus examination regularly. The examiners are blind. The progression of normal retinal vascularization and need to treatment will be documented and compared between the two study groups. The topical eye drops are used until the retinal vascularization are complete (45 week after LMP) or the patient needs to be treated.

ELIGIBILITY:
Inclusion Criteria:

* Premature infants who are candidate for retinopathy of prematurity (ROP) screening with ROP Type 2

Exclusion Criteria:

* Serious systemic problems
* Other ocular problems Except ROP

Max Age: 45 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 184 (Estimated)
Dates: Start 2019-06-02 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Stimulation of normal retinal vascularization and disease progression inhibition | 3 months
  Fundoscopy and examiner judgment which will be documented by retinal camera

SECONDARY OUTCOMES:
Any adverse event | 3 months
  Neonatologist and ophthalmologist examination

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmic Research Center, Tehran, Iran